CLINICAL TRIAL: NCT00006394
Title: Randomized Study of Growth Hormone on Bone Mineral Density in Patients With Adult Onset Growth Hormone Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Pennsylvania (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/15433; UPSM-209300; LILLY-B9R-US-GDEO
Record Dates: First submitted 2000-10-04; First posted 2000-10-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Osteoporosis; Growth Hormone Deficiency
Keywords: disease-related problem/condition; endocrine disorders; growth hormone deficiency; osteoporosis; quality of life; rare disease
MeSH Terms: conditions — Osteoporosis; Dwarfism, Pituitary; Endocrine System Diseases; Rare Diseases | interventions — Growth Hormone

INTERVENTIONS:
Drug: growth hormone

SUMMARY:
OBJECTIVES: I. Compare whether the bone tissue in the spine and hip improves in patients with adult onset growth hormone deficiency treated with growth hormone (GH) vs placebo.

II. Determine whether the blood samples of these patients show evidence of beneficial bone effects after treatment with GH.

III. Compare the quality of life of these patients treated with these 2 regimens.

IV. Determine the side effects of GH in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive growth hormone subcutaneously (SC) daily for 2 years. Arm II: Patients receive placebo SC daily for 2 years. Quality of life is assessed at the initial eligibility screening, then again within 1 month after the initial screening, and then at 1, 3, and 6 months during study therapy.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of adult onset growth hormone deficiency

--Patient Characteristics--

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 1997-04

CONTACTS AND LOCATIONS:
Overall Officials: Peter Snyder, Study Chair — University of Pennsylvania
Locations (7):
- United States (7):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Case Western Reserve University, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island